CLINICAL TRIAL: NCT04478734
Title: Multicentric Trial on the Use of Combined Therapy of Thiamine and Biotine in Patients With Huntington´s Disease
Brief Title: Trial of the Combined Use of Thiamine and Biotin in Patients With Huntington's Disease
Acronym: HUNTIAM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Collaborators: Ciberned (Centro de Investigación Biomédica en Red) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUNTIAM
Record Dates: First submitted 2020-02-11; First posted 2020-07-21 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-01

CONDITIONS: Huntington Disease
Keywords: thiamine and biotine; combination therapy
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Moderate doses (Experimental): moderate doses of combination therapy applying the minimum average dosage of thiamine and biotin used in patients with BTBGD
  Interventions: Drug: Moderate doses of Thiamine y Biotin
- High doses (Experimental): high doses of the combination therapy applying the average standard dosage of thiamine and biotin used in patients with BTBGD.
  Interventions: Drug: High doses of Thiamine y Biotin

INTERVENTIONS:
Drug: Moderate doses of Thiamine y Biotin — Thiamine 600 mg every day + Biotin 150mg every day
  Other Names: moderate doses of combination therapy
  Arms: Moderate doses
Drug: High doses of Thiamine y Biotin — Thiamine 1200 mg every day + Biotin 300mg every day
  Other Names: high doses of the combination therapy
  Arms: High doses

SUMMARY:
Evaluate the safety and tolerability of combined oral thiamine with biotin therapy in patients with Huntington´s disease in mild to moderate stages and it is intended to evaluate the biological effect of the treatment in the central nervous system of these patients using as the main biomarker the increase in the level of thiamine monophosphate (TMP) in cerebrospinal fluid (CSF) of these patients with Huntington Disease (HD) during a follow-up period of one year.

Our main hypothesis is that combined thiamine-biotin oral therapy is a secure and well-tolerated treatment, potentially capable of modifying the disease course or avoiding the progression of symptoms in early-stages HD patients

DETAILED DESCRIPTION:
The assessment of the safety and tolerability of the combined oral thiamine and biotin therapy in patients with HD will be performed by:

* Periodic clinical examination and anamnesis directed by a neurologist during face-to-face and non-contact visits.
* The collection of adverse effects during interviews of face-to-face visits to assess tolerability.
* Analytical monitoring with hematological and biochemical control (hepatic and renal function) during the dose escalation period, subsequently being this periodic control every 3 months, from signature of informed consent until the end the follow up.

The evaluation of the biological efficacy of treatment with combined oral thiamine and biotin therapy in increasing thiamine monophosphate (TMP) levels in cerebrospinal fluid (CSF) of patients with HD is to be performed by:

* The determination of thiamine levels: free thiamine, TMP, and thiamine pyrophosphate (TTP) in CSF and blood of patients at the beginning and after the end of the study.
* Comparison of thiamine levels (free, TMP and TTP) between the start and the end of the study in CSF and serum of patients with HD.

The evaluation of the biological efficacy of the treatment with combined oral thiamine and oral biotin therapy in neurodegeneration produced in HD will be performed by:

* Measurement of neurofilament light chain protein (NfL) levels in CSF at the baseline visit and after the end of the treatment.
* The obtained score in the motor and Total Functional Capacity (TFC) section of the Unified Huntington's Disease Rating Scale (UHDRS).
* Measurement of bradykinesia through quantitative motion measurement techniques (Quantitative motor assessment, Q-motor). Q-motor assessment relies on three-dimensional position sensors and pre-calibrated force translators, for standardized movement recording. This measurement will be made to patients in the pre-selection visit, randomization, and quarterly face-to-face visits.
* Score on the quality of life scale (SF-36).
* Variation in the overall clinical impression scale of the patient and the examiner.
* Measurement of the change in the volume of the caudate nucleus, white matter, and cortical thickness, as well as in the change of the Combined cerebral atrophy score. Measurements of cerebral structures will be acquired on magnetic resonance imaging scans (3T) at the baseline visit and after the end of the treatment.

To determine the sample size required to examine secondary and exploratory objectives, we based our estimations on the published thiamine-biotin treatment effects in preclinical HD models, and on the reported differences in CSF thiamine levels between HD patients and healthy subjects (Pico S, et al. 2021). According to the previous results, it is expected that a medium-to-high effect size (0.6 ≤ Cohen's d ≥ 0.8) would be necessary to restore TPP, TMP and Free-thiamine levels in CSF after treatment. Based on the parameter choices, for a desired power of 0.80 and a Type I error rate of 0.05, we estimate that we would need 24 HD patients to detect a standardized mean difference of 0.6. Sample size analysis was conducted using GPower 3.1.9.7 software.

The demographic data collection as well as the information related to all the variables analyzed during the study will be done through an electronic data collection notebook. The notification of adverse effects, severity, and relationship with study medication will be done through an electronic data collection notebook.

All statistical analyses will be conducted using SPSS v.26.0. IBM software and R studio software package. Linear regression will be used when the variables are quantitative (eg, scale measurements, CSF thiamine or NfL levels, among others) controlling for age, sex, CAG repetitions and motor symptom severity (UHDRS and UHDRS-Total Functional Capacity) at baseline as potential confounding variables. Logistic or multinomial regression when the variables are groups (binary or multinomial).

We will examine the association between the severity of disease and CSF thiamine among HD patients by fitting a linear mixed model for each clinical measurement, with age, sex, CAG repetitions and disease severity (UHDRS-TFC) as the covariates.

Magnetic resonance imaging performed during the study will be processed with specific neuroimaging programs for volumetry, diffusion and cortical thickness.

ELIGIBILITY:
Inclusion Criteria:

* Patients of legal age with manifest Huntington's disease with motor symptoms (chorea, dystonia or bradykinesia) and/or neuropsychiatric; and genetic confirmation of a number of repetitions of the cytosine-adenine-guanine trinucleotide (CAG triplet) in the HTT gene (coding for HTT) greater than or equal to 39
* Patients should be capable of giving informed consent and attending the planned visit of the study.
* Women of childbearing age should obtain a negative result in the serum or urine pregnancy test at the screening visit. They must also accept the use of appropriate contraceptive methods during the course of the clinical trial and men who have a partner of childbearing age, accept the use of contraceptive methods

Exclusion Criteria:

* Medical comorbidities considered clinically significant by the clinical judgment of the investigators.
* Pregnancy or lactation
* Patients with HD dependents on the basic routine daily life activities (UHDRS TFC < 7) or a severe cognitive decline.
* Active psychosis at the moment of the screening evaluation.
* Severe renal failure.
* Patients previously treated with thiamine and/or biotin or enrolled in other HD clinical trial with oligonucleotide antisense (IONIS-HTTRX (RG6042).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed by clinical examination anamnesis and Analytical monitoring with hematological and biochemical control (hepatic and renal function) | From signature of informed consent form, at all scheduled visits, to end of follow up week 52
  Patient´s condition and emergence of comorbidity by clinical examination and anamnesis directed by a neurologist, by measuring of vital signs (blood pressure, heart rate,breath rate weight and height)

SECONDARY OUTCOMES:
The evaluation of the efficacy of treatment with combined oral thiamine and biotin therapy in increasing thiamine monophosphate (TMP) levels in CSF of patients with HD | At baseline (week 0) and visit 8 (week 48)
  Determination and comparison of thiamine levels (free, TMP and TTP) in CSF and blood at the beginning and the end of the treatment.

OTHER OUTCOMES:
Evaluate the biological effect of the combined thiamine-biotin oral therapy in the neurodegeration of HD patients | At baseline (week 0) and visit 8 (week 48)
  Measurement of the change in CSF NfL levels of patients with HD treated with the combined thiamine-biotin therapy
Evaluate the biological effect of the combined thiamine-biotin oral therapy in the neuroimaging progression markers in patients with HD | At baseline (week 0) and visit 8 (week 48)
  Measurement of the change in the volume of the caudate nucleus, white matter and cortical thickness, as well as in the combined cerebral atrophy score; comparing these values with those described in prospective registries of patients with HD.
Evaluate the effect of the combined thiamine-biotin oral therapy in the quality of life of patients with HD | At baseline (week 0), week 24 and week 48
  Changes in the 36-Item Short Form Health Survey (SF-36) score of the quality of life. Short Form 36 Health Survey (SF-36 ) consists of 35 punctually items, divided into 8 dimensions: Physical Function, Physical Role, Emotional Role, Social Function, Mental Health, General Health, Body Pain and Vitality. It also contains an additional item that is not part of any dimension and that measures the change in health over time. The scores of the 8 dimensions of SF-36 are arranged in such a way that the higher the value recorded, the better the corresponding health status. scale (SF-36).
Evaluate the clinical effect of the combined thiamine-biotin oral therapy in the severity of motor symptoms of patients with HD | At baseline (week 0), week 24 and week 48
  Evaluate changes in the score of the UHDRS motor scale and UHDRS- Total functional capacity.
Evaluate the clinical effect of the combined thiamine-biotin oral therapy in the severity of bradykinesia of patients with HD. | At baseline (week 0), week 12, week 24, week 36 and week 48
  Evaluate changes in the score of Quantitative-motor assessments (Q-motor). Measurement of bradykinesia will be done through quantitative movement measurement techniques.
Evaluate the effect of the combined thiamine-biotin oral therapy in the global severity of disease of patients with HD | At baseline (week 0), week 24 and week 48
  Changes in the score of The Clinical Global Impressions - Severity scale-S (CGI-C).
  The CGI provides a brief of the patient's global functioning prior to and after initiating a study medication.
  Comprises two measures evaluating the following: (a) severity of psychopathology from 1 to 7 and (b) change from the initiation of treatment on a similar seven-point scale. CGI-C scores range from 1 (very much improved) through to 7 (very much worse).

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Mir Rivera, MD/PhD, Study Director — Institute of Biomedicine of Seville (IBiS); Clara M. Rosso Fernández, Principal Investigator — Virgen del Rocío University Hospital Research and Clinical Trials Unit
Locations (3):
- Spain (3):
  - Hospital Universitario de San Sebastián, San Sebastián, San Sebastian
  - Virgen del Rocío Hospital, Seville, Seville
  - Hospital Ramón y Cajal, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Once the study is completed and the data processed, the results will be shared
Supporting Information: Study Protocol, CSR
Time Frame: After the primary completion date and submit results information
Access Criteria: collaborating researchers